CLINICAL TRIAL: NCT03958552
Title: Palliative Care Consultations for Persons in the Medicare Skilled Nursing Facility (SNF) Setting
Brief Title: Palliative Care Consultations in the Skilled Nursing Facility (SNF) Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Joan Carpenter, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00099506
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Palliative Care; Advance Care Planning; Skilled Nursing Facilities
Keywords: Palliative Care Consultation; Medicare; Skilled Nursing

STUDY DESIGN:
Intervention Model Description: Pre-post design where control data will be collected prior to intervention being implemented
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants will receive the standard Medicare Skilled Nursing Facility care.
- Palliative Care Consult (Experimental): Participants will receive the standard Medicare Skilled Nursing Facility care plus a Palliative Care Consultation with a trained provider.
  Interventions: Other: Palliative Care Consultation

INTERVENTIONS:
Other: Palliative Care Consultation — Trained provider will discuss illness trajectories, establish and communicate patient-directed goals that guide health care decisions, identify and treat illness-related symptoms, and identify psycho-spiritual needs and approaches to mitigate suffering.
  Arms: Palliative Care Consult

SUMMARY:
Close to one-third of Medicare decedents use the Medicare skilled nursing facility (SNF) benefit in the 6 months prior to death. SNF care often increases the risk for more aggressive, potentially burdensome treatments and unrecognized or undertreated symptoms. Palliative care is goal-directed, patient and family-centered care that focuses on a wide range of physical, psychosocial, and spiritual needs for persons with serious, life-limiting illnesses. Effective palliative care relieves suffering, enhances communication, and improves end-of-life care and decision making for seriously ill older adults. Despite its association with improved quality of care, higher satisfaction, and better symptom management at the end of life, palliative care is not widely available to Medicare patients in the Skilled Nursing Facility (SNF) setting. Palliative care consultation (PCC) is one approach that can potentially improve care for older adults with advanced illness in SNFs. This pilot study will test an evidence-based palliative care consult intervention for older adult SNF patients in nursing homes by comparing the patient/family caregiver reported quality of life in two participant groups: one receiving a PCC and the other receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a participating nursing home under the Medicare SNF benefit
* English speaking
* If non-verbal or unable to participate in a conversation, a legally authorized representative(LAR) or surrogate decision maker who can participate in the study
* A diagnosis of one or more advanced serious illness using established criteria
* One global indicator for a PCC at SNF admission (i.e., primary provider would not be surprised if patient died in 12 months; frequent hospital or SNF admissions; complex care requirements; decline in function; feeding intolerance; or unintended decline in weight)

Exclusion Criteria:

* Patients who have previously received or are referred for a SNF-based PCC by their primary care team

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Carpenter, PhD, Principal Investigator — UMSON
Locations (1):
- Acts Continuing Care Retirement Communities, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared per an agreement between UPenn and participating SNFs

REFERENCES:
- [Background] Aragon K, Covinsky K, Miao Y, Boscardin WJ, Flint L, Smith AK. Use of the Medicare posthospitalization skilled nursing benefit in the last 6 months of life. Arch Intern Med. 2012 Nov 12;172(20):1573-9. doi: 10.1001/archinternmed.2012.4451. PMID 23026981
- [Background] Retrum JH, Gozansky WS, Lahoff DG, Rosenberg EL, Tropeano LE, Owens BA, Fischer SM. A Need for More Palliative Focused Care: A Survey of Colorado Skilled Care Facilities. J Am Med Dir Assoc. 2015 Aug 1;16(8):712-3. doi: 10.1016/j.jamda.2015.05.011. Epub 2015 Jul 6. No abstract available. PMID 26159824
- [Background] Carpenter JG, Berry PH, Ersek M. Nursing home care trajectories for older adults following in-hospital palliative care consultation. Geriatr Nurs. 2017 Nov-Dec;38(6):531-536. doi: 10.1016/j.gerinurse.2017.03.016. Epub 2017 Apr 28. PMID 28457493
- [Background] Givens JL, Mitchell SL, Kuo S, Gozalo P, Mor V, Teno J. Skilled nursing facility admissions of nursing home residents with advanced dementia. J Am Geriatr Soc. 2013 Oct;61(10):1645-50. doi: 10.1111/jgs.12476. Epub 2013 Oct 1. PMID 24117283
- [Background] Miller SC, Lima JC, Looze J, Mitchell SL. Dying in U.S. nursing homes with advanced dementia: how does health care use differ for residents with, versus without, end-of-life Medicare skilled nursing facility care? J Palliat Med. 2012 Jan;15(1):43-50. doi: 10.1089/jpm.2011.0210. Epub 2011 Dec 16. PMID 22175816
- [Background] Mor V, Intrator O, Feng Z, Grabowski DC. The revolving door of rehospitalization from skilled nursing facilities. Health Aff (Millwood). 2010 Jan-Feb;29(1):57-64. doi: 10.1377/hlthaff.2009.0629. PMID 20048361
- [Background] Boockvar K, Fishman E, Kyriacou CK, Monias A, Gavi S, Cortes T. Adverse events due to discontinuations in drug use and dose changes in patients transferred between acute and long-term care facilities. Arch Intern Med. 2004 Mar 8;164(5):545-50. doi: 10.1001/archinte.164.5.545. PMID 15006832
- [Background] Murray LM, Laditka SB. Care transitions by older adults from nursing homes to hospitals: implications for long-term care practice, geriatrics education, and research. J Am Med Dir Assoc. 2010 May;11(4):231-8. doi: 10.1016/j.jamda.2009.09.007. Epub 2010 Mar 24. PMID 20439041
- [Background] Boockvar KS, Gruber-Baldini AL, Burton L, Zimmerman S, May C, Magaziner J. Outcomes of infection in nursing home residents with and without early hospital transfer. J Am Geriatr Soc. 2005 Apr;53(4):590-6. doi: 10.1111/j.1532-5415.2005.53205.x. PMID 15817003
- [Background] Miller SC, Lima JC, Intrator O, Martin E, Bull J, Hanson LC. Palliative Care Consultations in Nursing Homes and Reductions in Acute Care Use and Potentially Burdensome End-of-Life Transitions. J Am Geriatr Soc. 2016 Nov;64(11):2280-2287. doi: 10.1111/jgs.14469. Epub 2016 Sep 19. PMID 27641157
- [Background] Miller SC, Dahal R, Lima JC, Intrator O, Martin E, Bull J, Hanson LC. Palliative Care Consultations in Nursing Homes and End-of-Life Hospitalizations. J Pain Symptom Manage. 2016 Dec;52(6):878-883. doi: 10.1016/j.jpainsymman.2016.05.017. Epub 2016 Sep 17. PMID 27650008
- [Background] Huskamp HA, Kaufmann C, Stevenson DG. The intersection of long-term care and end-of-life care. Med Care Res Rev. 2012 Feb;69(1):3-44. doi: 10.1177/1077558711418518. Epub 2011 Sep 8. PMID 21903662
- [Background] Ersek M, Carpenter JG. Geriatric palliative care in long-term care settings with a focus on nursing homes. J Palliat Med. 2013 Oct;16(10):1180-7. doi: 10.1089/jpm.2013.9474. Epub 2013 Aug 28. PMID 23984636
- See also: The National Consensus Project for Quality Palliative Care. Clinical Practice Guidelines for Quality Palliative Care, 3rd edition — https://www.nationalcoalitionhpc.org/ncp/

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care (Control): Participants received the standard Medicare Skilled Nursing Facility care, Patient Outcome Survey (POS) at enrollment and follow-up 15-21 days later.
- Palliative Care Consult: Participants received the standard Medicare Skilled Nursing Facility care plus a Palliative Care Consultation. They also received a Patient Outcome Survey (POS) at enrollment and followup POS and Consultation Satisfaction Questionnaire (CSQ) 15-21 later.
Period: Overall Study
Arm/Group | Standard Care (Control) | Palliative Care Consult
Started | 10 | 35
Completed | 10 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Care: Participants received the standard Medicare Skilled Nursing Facility care.
- Palliative Care Consult: Participants received the standard Medicare Skilled Nursing Facility care plus a Palliative Care Consultation with a trained provider.
  Palliative Care Consultation: Trained provider discussed illness trajectories, establish and communicate patient-directed goals that guide health care decisions, identify and treat illness-related symptoms, and identify psycho-spiritual needs and approaches to mitigate suffering.
- Total: Total of all reporting groups
Arm/Group | Standard Care | Palliative Care Consult | Total
Number analyzed (Participants) | 10 | 35 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 35 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 27 | 34
  Male | 3 | 8 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 35 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 34 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 35 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Patient Quality of Life Surveys
Description: The Patient Outcome Survey (POS) 10 item Survey that measures quality of life in five dimensions: 1) physical; 2) emotional; 3) psychological; 4) spiritual needs, and 5) provision of information and support. Items scored on a 5 point Likert Scale (0=not at all, 4= overwhelmingly) based on symptom/need in the past week. Overall profile score is calculated by summing responses (range 0-40). Higher values represent a worse outcome.
Time Frame: Collected upon admission to the nursing home and enrollment and again 15-21 days after enrollment in the study (control group) or intervention received (intervention group).
Population: Both intervention and control groups are administered a baseline POS and follow up POS.
Measure: Number; unit: participants
Groups:
- Standard Care (Control Group): Participants received the standard Medicare Skilled Nursing Facility care.
- Palliative Care Consult (Intervention Group): Participants received the standard Medicare Skilled Nursing Facility care plus a Palliative Care Consultation with a trained provider.
  Palliative Care Consultation: Trained provider discussed illness trajectories, establish and communicate patient-directed goals that guide health care decisions, identify and treat illness-related symptoms, and identify psycho-spiritual needs and approaches to mitigate suffering.
Arm/Group | Standard Care (Control Group) | Palliative Care Consult (Intervention Group)
Number analyzed (Participants) | 10 | 35
participants
  Completed Baseline POS | 10 | 35
  Completed Follow up POS | 10 | 35

2. Secondary Outcome: Number of Participants Who Completed the Consult Satisfaction Survey (CSQ)
Description: Measured using the Consultation Satisfaction Questionnaire (CSQ). The CSQ is an 18 item patient/caregiver-reported instrument that measures communication and satisfaction of a consult in four domains: 1) general satisfaction, 2) professional care, 3) depth of relationship, 4) perceived length of consultation.(scale format: 5-point Likert Scale (0= strongly disagree, 4=strongly agree).Overall score is calculated by summing responses (range 0-72). Higher values represent a worse outcome.
Time Frame: Collected within 15-21days of palliative care consultation for the intervention group.
Population: Participants in the Control arm were not administered the CSQ survey. Only participants in the intervention group were administered the CSQ survey
Measure: Number; unit: participants
Groups:
- Standard Care (Control): Participants received the standard Medicare Skilled Nursing Facility care.
- Palliative Care Consult (Intervention): Participants received the standard Medicare Skilled Nursing Facility care plus a Palliative Care Consultation with a trained provider.
Arm/Group | Standard Care (Control) | Palliative Care Consult (Intervention)
Number analyzed (Participants) | 0 | 10
participants |  | 10

3. Secondary Outcome: Adherence to SNF-PCC Recommendations
Description: Adherence Protocol. Medical record review and/or phone interview with patient/caregiver
  We will determine a recommendation adherence score after each participants' SNF-PCC. Each recommendation will be assigned 2 points, then we will define full (2 points), partial (1 point) and no adherence (0 point) to each recommendation. We will sum the points for each SNF-PCC recommendation and use this as the denominator. We will sum each recommendation with full, partial, no adherence and use this as the numerator. The fraction will be converted to a percentage ranging from 0-100% reflecting the recommendation adherence score.
Time Frame: 30 Days post-admission
Population: Data were not collected due to study teams limited access to the medical records to review Adherence to SNF-PCC recommendations (due to Covid 19)
Arm/Group | Standard Care (Control Group) | Palliative Care Consult (Intervention)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 21 days
Arm/Group | Standard Care | Palliative Care Consult
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/35
Other Adverse Events (participants affected / at risk) | 0/10 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT03958552/Prot_SAP_000.pdf